CLINICAL TRIAL: NCT02447120
Title: Topcon 3D OCT-1 Maestro Reference Database Study II
Status: Completed | Type: Observational
Sponsor: Topcon Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Organization: Topcon Corporation (Industry)
Other Study IDs: Maestro_NDB_II
Record Dates: First submitted 2015-05-12; First posted 2015-05-18 (Estimated); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Healthy
Keywords: Volunteers with Healthy Eyes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normal Eyes: Subjects with no known ocular diseases will be scanned with the Maestro device
  Interventions: Device: 3D OCT-1 Maestro

INTERVENTIONS:
Device: 3D OCT-1 Maestro — OCT machines used for diagnostic purposes

SUMMARY:
The objective of this study is to collect OCT measurement data on normal healthy eyes in order to determine the reference limits for Topcon 3D OCT-1 Maestro based on the percentile points for 1%, 5%, 95%, and 99%.

DETAILED DESCRIPTION:
The objective of this study is to collect OCT measurement data on normal healthy eyes in order to determine the reference limits for Topcon 3D OCT-1 Maestro based on the percentile points for 1%, 5%, 95%, and 99%.

ELIGIBILITY:
Inclusion Criteria for Normal Group

1. Subjects 18 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. Subjects presenting at the site with normal eyes (eyes without pathology)
4. lOP <= 21 mmHg bilaterally
5. BCVA 20/40 or better (each eye)
6. Both eyes must be free of eye disease

Exclusion Criteria for Normal Group

1. Subjects previously enrolled in either the Maestro AP study or the Maestro2 study
2. Subjects unable to tolerate ophthalmic imaging
3. Subject with ocular media not sufficiently clear to obtain acceptable OCT images
4. HFA visual field (24-2 Sita Standard, white on white) result unreliable (based on manufacturer's recommendation), defined as fixation losses > 20% or false positives> 33%, or false negatives> 33%
5. Visual field defects consistent with glaucomatous optic nerve damage based on with at least one of the following two findings:

   * On pattern deviation (PD), there exists a cluster of 3 or more points in an expected location of the visual field depressed below the 5% level, at least 1 of which is depressed below the 1% level;
   * Glaucoma hemi-field test "outside normal limits."
6. Presence of any ocular pathology except for cataract
7. Narrow angle
8. History of leukemia, dementia or multiple sclerosis
9. Concomitant use of hydroxychloroquine and chloroquine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects without eye disease
Sampling Method: Non-Probability Sample
Enrollment: 504 (Actual)
Dates: Start 2015-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Retinal Thickness | 1 minute

CONTACTS AND LOCATIONS:
Overall Officials: Charles Reisman, MS, Study Chair — Topcon Corporation
Locations (7):
- United States (7):
  - UAB School of Optometry, Birmingham, Alabama
  - Southern California College of Optometry, Fullerton, California
  - Valley Eyecare Center, Livermore, California
  - Western University of Health Sciences, Pomona, California
  - Illinois College of Optometry, Chicago, Illinois
  - New York VA, Jamaica, New York
  - SUNY College of Optometry, New York, New York